CLINICAL TRIAL: NCT00325897
Title: Effect of Chronic Macrolide Administration on the Frequency and Severity of COPD Exacerbations
Brief Title: Macrolide Azithromycin to Prevent Rapid Worsening of Symptoms Associated With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 0510M76766; U10HL074424-03 (NIH)
Record Dates: First submitted 2006-05-12; First posted 2006-05-15 (Estimated); Results first posted 2012-06-07 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Macrolides; Azithromycin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azithromycin, 250 mg (Active Comparator): Macrolide Antibiotic (Azithromycin)
  Interventions: Drug: Macrolide Antibiotic (Azithromycin)
- Placebo (Placebo Comparator): Inactive
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Macrolide Antibiotic (Azithromycin) — Azithromycin (daily capsule, 250 mg for 12 months)
  Other Names: Zithromax; Zmax
  Arms: Azithromycin, 250 mg
Drug: Placebo — Placebo taken on a daily basis
  Other Names: sugar pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if long-term administration of a macrolide antibiotic will reduce worsening of symptoms among individuals with chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
BACKGROUND:

The prevalence, morbidity, mortality, and treatment cost of COPD are high and increasing. COPD is the sixth leading cause of death worldwide and is the only condition in the top 10 causes of death that has an increasing prevalence and mortality. The cost of health care for patients with COPD in the U.S. is approximately $6.5 billion per year; acute exacerbations account for between 31% and 68% of that cost. Macrolide antibiotics may reduce the frequency and/or severity of COPD exacerbations, as a result of their antibacterial properties and anti-inflammatory effects. Long-term administration of macrolide antibiotics in patients with a number of other pulmonary disorders has resulted in clinically important improvements. It is hypothesized that administration of a macrolide antibiotic (azithromycin) for 1 year, when added to usual care, will decrease the frequency and severity of COPD exacerbations. If this hypothesis is correct, the proposed treatment is also expected to reduce the mortality of COPD patients.

DESIGN NARRATIVE:

This is a prospective, randomized, double-blind, placebo-controlled study that will enroll 1130 patients with at least moderately severe COPD who, based on clinical indicators, have an increased likelihood of experiencing an acute exacerbation during the study period. Patients will be monitored monthly, including careful assessments of possible macrolide-related side effects. The exclusion criteria for this study will include a variety of conditions or medications that are known to adversely interact with macrolides. The primary endpoint of this study is time until the first acute COPD exacerbation. The secondary endpoints include macrolide-related side effects, the incidence of macrolide-resistant bacterial colonization, quality of life, and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of at least moderate Chronic Obstructive Pulmonary Disease (COPD), as defined by the following Global Initiative for COPD (GOLD) criteria:

  1. Post-bronchodilator forced expiratory volume in one second (FEV1)/forced vital capacity (FVC) ratio of less than 70%
  2. Post-bronchodilator FEV1 less than 80% predicted, with or without chronic symptoms
* Cigarette consumption of 10 pack-years or more (may or may not be active smokers)
* Meets one or more of the following four conditions:

  1. Current, or history of, supplemental O2 use
  2. Received a course of systemic corticosteroids for respiratory problems within 1 year prior to study entry
  3. Visited an emergency department for a COPD exacerbation within 1 year prior to study entry
  4. Hospitalized for a COPD exacerbation within 1 year prior to study entry
* Willing to make return visits
* Available by telephone for duration of study
* Minimum of 4 weeks from the most recent acute exacerbation (have not received a course of systemic corticosteroids, an increased dose of chronically administered systemic corticosteroids, and/or antibiotics for an acute exacerbation for a minimum of 4 weeks from the time of study entry)

Exclusion Criteria:

* Diagnosis of asthma
* Diagnosis other than COPD that results in the patient being either medically unstable, or having a predicted life expectancy less than 3 years
* Special patient groups (i.e., prisoners, pregnant women, or institutionalized patients)
* Women who are at risk of becoming pregnant during the study (pre-menopausal) and who refuse to use acceptable birth control (i.e., hormone-based oral or barrier contraceptive) for the duration of the study
* History of hypersensitivity to any macrolide antibiotic
* Taking any of the following medications:

  1. Cisapride
  2. Ergot derivatives
  3. Pimozide
  4. Disopyramide
  5. Cyclosporin
  6. Tacrolimus
  7. Nelfinavir
  8. Bromocriptine
  9. Hexobarbital
* Corrected QT interval (QTc) on electrocardiogram exceeding 440 ms
* Taking rifabutin or rifampin
* Chronic hepatic insufficiency
* Chronic renal insufficiency
* Diagnosis of bronchiectasis (defined as production of greater than one-half cup of purulent sputum/day)
* If, for either ear, formal audiometric testing in a sound booth results in a pure tone average (i.e., the average of the thresholds for the 4 frequencies 1000, 2000, 3000, or 4000) exceeding 50 decibel (dB), or if the threshold at any one frequency exceeds 60 dB, then the participant will be counseled by the audiologist concerning hearing aids and/or referral to an otolaryngologist. In addition, the audiologist may discuss with the participant whether or not to continue in the study. Following the examination and counseling, the participant will also discuss whether or not to continue in the study with one of the study investigators. If it is found that a participant's pure tone average in the two ears differs by more than 15 dB, or if the difference in the two ears for any one frequency exceeds 20 dB, then the participant will not be eligible for randomization into the study unless cleared by an otolaryngologist

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1142 (Actual)
Dates: Start 2006-03; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard K. Albert, MD, Principal Investigator — Denver City-County Health/Hospitals Department; William C. Bailey, MD, Principal Investigator — University of Alabama at Birmingham; Richard Casaburi, MD, PhD, Principal Investigator — Harbor-UCLA Research & Education Institute; John E. Connett, PhD, Principal Investigator — University of Minnesota; Gerard J. Criner, MD, Principal Investigator — Temple University; Stephen C. Lazarus, MD, Principal Investigator — University of California at San Francisco; Fernando J. Martinez, MD, Principal Investigator — University of Michigan; Dennis E. Niewoehner, MD, Principal Investigator — Minnesota Veterans Medical Research and Education Foundation; John J. Reilly, MD, Principal Investigator — Brigham and Women's Hospital; Steven M. Scharf, MD, PhD, Principal Investigator — University of Maryland, Baltimore; Frank Sciurba, MD, Principal Investigator — University of Pittsburgh
Locations (10):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California at San Francisco, San Francisco, California
  - Harbor-UCLA Research & Education Inst., Torrance, California
  - Denver City-County Health/Hospitals Dept., Denver, Colorado
  - University of Maryland Baltimore, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Minnesota Veterans Research Inst., Minneapolis, Minnesota
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Camac ER, Voelker H, Criner GJ; COPD Clinical Research Network and the Canadian Institutes of Health Research. Impact of COPD exacerbations leading to hospitalization on general and disease-specific quality of life. Respir Med. 2021 Sep;186:106526. doi: 10.1016/j.rmed.2021.106526. Epub 2021 Jun 29. PMID 34229290
- [Derived] Leitao Filho FS, Ra SW, Mattman A, Schellenberg RS, Criner GJ, Woodruff PG, Lazarus SC, Albert R, Connett JE, Han MK, Martinez FJ, Leung JM, Paul Man SF, Aaron SD, Reed RM, Sin DD; Canadian Respiratory Research Network (CRRN). Serum IgG subclass levels and risk of exacerbations and hospitalizations in patients with COPD. Respir Res. 2018 Feb 14;19(1):30. doi: 10.1186/s12931-018-0733-z. PMID 29444682
- [Derived] Brown KE, Sin DD, Voelker H, Connett JE, Niewoehner DE, Kunisaki KM; COPD Clinical Research Network. Serum bilirubin and the risk of chronic obstructive pulmonary disease exacerbations. Respir Res. 2017 Oct 24;18(1):179. doi: 10.1186/s12931-017-0664-0. PMID 29065885
- [Derived] Wetherbee EE, Niewoehner DE, Sisson JH, Lindberg SM, Connett JE, Kunisaki KM. Self-reported alcohol intake and risk of acute exacerbations of chronic obstructive pulmonary disease: a prospective cohort study. Int J Chron Obstruct Pulmon Dis. 2015 Jul 20;10:1363-70. doi: 10.2147/COPD.S86572. eCollection 2015. PMID 26229455
- [Derived] Geiger-Brown J, Lindberg S, Krachman S, McEvoy CE, Criner GJ, Connett JE, Albert RK, Scharf SM. Self-reported sleep quality and acute exacerbations of chronic obstructive pulmonary disease. Int J Chron Obstruct Pulmon Dis. 2015 Feb 20;10:389-97. doi: 10.2147/COPD.S75840. eCollection 2015. PMID 25759571
- [Derived] Han MK, Tayob N, Murray S, Dransfield MT, Washko G, Scanlon PD, Criner GJ, Casaburi R, Connett J, Lazarus SC, Albert R, Woodruff P, Martinez FJ. Predictors of chronic obstructive pulmonary disease exacerbation reduction in response to daily azithromycin therapy. Am J Respir Crit Care Med. 2014 Jun 15;189(12):1503-8. doi: 10.1164/rccm.201402-0207OC. PMID 24779680
- [Derived] Albert RK, Connett J, Curtis JL, Martinez FJ, Han MK, Lazarus SC, Woodruff PG. Mannose-binding lectin deficiency and acute exacerbations of chronic obstructive pulmonary disease. Int J Chron Obstruct Pulmon Dis. 2012;7:767-77. doi: 10.2147/COPD.S33714. Epub 2012 Nov 23. PMID 23226013
- [Derived] Albert RK, Connett J, Bailey WC, Casaburi R, Cooper JA Jr, Criner GJ, Curtis JL, Dransfield MT, Han MK, Lazarus SC, Make B, Marchetti N, Martinez FJ, Madinger NE, McEvoy C, Niewoehner DE, Porsasz J, Price CS, Reilly J, Scanlon PD, Sciurba FC, Scharf SM, Washko GR, Woodruff PG, Anthonisen NR; COPD Clinical Research Network. Azithromycin for prevention of exacerbations of COPD. N Engl J Med. 2011 Aug 25;365(8):689-98. doi: 10.1056/NEJMoa1104623. PMID 21864166
- [Derived] Kunisaki KM, Niewoehner DE. Antibiotic prophylaxis for chronic obstructive pulmonary disease: resurrecting an old idea. Am J Respir Crit Care Med. 2008 Dec 1;178(11):1098-9. doi: 10.1164/rccm.200808-1315ED. No abstract available. PMID 19023036
- See also: Published manuscript reporting main results — https://www.ncbi.nlm.nih.gov/pubmed/21864166

RESULTS

PARTICIPANT FLOW:
Groups:
- Azithromycin: Azithromycin, 250 mg
- Placebo: Inactive sugar pill
Period: Overall Study
Arm/Group | Azithromycin | Placebo
Started | 570 | 572
Completed | 558 | 559
Not Completed | 12 | 13
Not completed — Lost to Follow-up | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin | Placebo | Total
Number analyzed (Participants) | 570 | 572 | 1142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 277 | 261 | 538
  >=65 years | 293 | 311 | 604
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (8.7) | 65.5 (8.4) | 65.1 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 234 | 229 | 463
  Male | 336 | 343 | 679
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 14 | 25
  Not Hispanic or Latino | 559 | 558 | 1117
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — All applicable categories were checked for each participant.
  Participants
    American Indian or Alaska Native | 2 | 2 | 4
    Asian | 6 | 4 | 10
    Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
    Black or African American | 79 | 89 | 168
    White | 463 | 457 | 920
    More than one race | 20 | 18 | 38
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 570 | 572 | 1142

OUTCOME MEASURES:

1. Primary Outcome: Time Until First Occurrence of Acute Chronic Obstructive Pulmonary Disease (COPD) Exacerbation
Description: Time until first occurrence of acute Chronic Obstructive Pulmonary Disease (COPD) exacerbation. Acute exacerbations are defined as a "complex of respiratory symptoms (increase or new onset) of more than one of the following: cough, sputum, wheezing, dyspnea, or chest tightness with a duration of at least three days requiring treatment with antibiotics and/or systemic steroids "
Time Frame: Measured monthly through 13 months
Population: Participants that had any follow-up data were included in analysis.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Azithromycin: Azithromycin 250 mg
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 558 | 559
Days | 266 [227 to 313] | 174 [143 to 215]

2. Secondary Outcome: Exacerbations/Patient Year
Description: Acute exacerbations are defined as a "complex of respiratory symptoms (increase or new onset) of more than one of the following: cough, sputum, wheezing, dyspnea, or chest tightness with a duration of at least three days requiring treatment with antibiotics and/or systemic steroids "
Time Frame: Measured monthly until 13 months
Population: Participants with any follow-up data were analyzed.
Measure: Number; unit: exacerbations/patient year
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 558 | 559
exacerbations/patient year | 1.48 | 1.83

3. Secondary Outcome: Number of Emergency Department Visits as a Result of Acute Exacerbations
Time Frame: Measured monthly for 12 months
Measure: Number; unit: Visits
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 570 | 572
Visits | 199 | 257

4. Secondary Outcome: Number of Hospital Admissions as a Result of Acute Exacerbations
Time Frame: Measured monthly for 12 months
Measure: Number; unit: Hospitalizations
Arm/Group | Azithromycin | Placebo
Number analyzed (Participants) | 570 | 572
Hospitalizations | 156 | 200

5. Secondary Outcome: Change in Age-adjusted Hearing Threshold
Description: Assessed by audiometry for four sound frequencies (1000, 2000, 3000, 4000 Hz). The maximum was computed for each threshold in each ear for all frequencies, then the differences between visits were assessed.
Time Frame: Baseline and 12 months
Population: Participants with both baseline and one-year audiometry data available were analyzed.
Measure: Mean (Standard Deviation); unit: Decibels (db)
Arm/Group | Azithromycin, 250 mg | Placebo
Number analyzed (Participants) | 420 | 426
Decibels (db) | -1.2 (4.2) | -0.9 (4.1)

6. Secondary Outcome: Incidence of Macrolide-resistant Bacterial Colonization of the Nasopharynx or Sputum
Description: Cultures from 68% of the participants in the azithromycin group and 70% in the placebo group who were not colonized with selected respiratory pathogens at the time of enrollment but who became colonized during the course of the study were available for susceptibility testing for the incidence of macrolide-resistant bacterial colonization.
Time Frame: Baseline
Population: Using cultures from participants who were not colonized with selected respiratory pathogens at the time of enrollment but who became colonized during the course of the study, samples were available from 68% of the participants in the azithromycin group and 70% in the placebo group among these cultures.
Measure: Number; unit: Participants
Arm/Group | Azithromycin, 250 mg | Placebo
Number analyzed (Participants) | 44 | 49
Participants | 23 | 28

7. Secondary Outcome: Incidence of Macrolide-resistant Bacterial Colonization of the Nasopharynx or Sputum
Description: Cultures from some participants who were not colonized with selected respiratory pathogens at the time of enrollment but who became colonized during the course of the study were available for susceptibility testing for the incidence of macrolide-resistant bacterial colonization.
Time Frame: During Course of Study (either month 3, 6, 9, or 12)
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | Azithromycin, 250 mg | Placebo
Number analyzed (Participants) | 47 | 108
participants | 38 | 44

ADVERSE EVENTS:
Time Frame: 13 months
Arm/Group | Azithromycin | Placebo
Serious Adverse Events (participants affected / at risk) | 217/570 | 217/572
Other Adverse Events (participants affected / at risk) | 500/570 | 444/572
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azithromycin (N=570) | Placebo (N=572)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 24 (26) | 37 (41)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (7) | 8 (13)
Digestive (Gastrointestinal disorders) | 15 (15) | 18 (21)
Circulatory (Cardiac disorders) | 32 (32) | 31 (36)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 120 (145) | 109 (170)
Other (General disorders) | 100 (113) | 101 (114)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azithromycin (N=570) | Placebo (N=572)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 7 (13) | 24 (27)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (13) | 15 (16)
Digestive (Gastrointestinal disorders) | 62 (89) | 78 (104)
Circulatory (Cardiac disorders) | 34 (49) | 29 (42)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 185 (566) | 244 (657)
Other (General disorders) | 319 (1132) | 331 (1176)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No